CLINICAL TRIAL: NCT00472966
Title: Open Label Study to Evaluate the Efficacy and Safety of Sequential Therapy With Fluocinolone Acetonide 0.01%, Hydroquinone (HQ) 4% and Tretinoin 0.05% (TriLuma® Cream) and a Series of Glycolic Acid Peels for the Treatment of Melasma
Brief Title: Efficacy and Safety of Therapy With Tri-Luma® Cream in Sequence With Glycolic Acid Peels for Melasma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Ronald W. Gottschalk, MD / Medical Director, Galderma Laboratories, L.P.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US10031
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2008-03

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Fluocinolone Acetonide; hydroquinone; Tretinoin; Base Sequence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Fluocinolone acetonide 0.1%/hydroquinone 4%/tretinoin 0.05% Cream in sequence with glycolic acid peels
  Interventions: Drug: Fluocinolone acetonide 0.1%/hydroquinone 4%/tretinoin 0.05% Cream in sequence with glycolic acid peels

INTERVENTIONS:
Drug: Fluocinolone acetonide 0.1%/hydroquinone 4%/tretinoin 0.05% Cream in sequence with glycolic acid peels — Apply cream once daily at night. Subjects will be asked to discontinue use of Fluocinolone acetonide/hydroquinone/tretinoin Cream 2 days prior to the peel and restart 2 days after the peel; Glycolic Acid Peels - In office treatment at weeks 2, 4, 6, 8 and 10
  Other Names: Tri-Luma® Cream; NeoStrata® Glycolic Acid Skin Renewal Peel

SUMMARY:
To determine the effectiveness and safety of sequential therapy with of Tri-Luma® Cream and a series of Glycolic Acid peels in treatment of moderate to severe melasma.

DETAILED DESCRIPTION:
To determine the efficacy and safety of sequential therapy with Fluocinolone acetonide 0.01%, Hydroquinone 4% and Tretinoin 0.05%, and a series of Glycolic Acid peels in the treatment of moderate to severe melasma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with moderate to severe melasma

Exclusion Criteria:

* Subjects under treatment for a dermatologic condition, which may interfere with the safe evaluation of the study combination (e.g. eczema, psoriasis, severe sun-damage, dermatitis)
* Subjects with a diagnosis of skin cancer (BCE, SCC, Melanoma) in the areas to be treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Efficacy - Improvement in Investigator's global assessment of melasma | 12 weeks

SECONDARY OUTCOMES:
Safety - Tolerability assessments and adverse event reporting | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (1):
- Skin Care Research, Inc., Boca Raton, Florida, United States